CLINICAL TRIAL: NCT07048106
Title: Natural History and Structural Consequences of a Diseased Bruch's Membrane in Pseudoxanthoma Elasticum (PXE)
Brief Title: Progression Assessment of PXE-associated Alterations
Acronym: PAPA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Kristina Pfau, Principal Investigator, University Hospital, Bonn
Other Study IDs: UBonn
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pseudoxanthoma Elasticum; Angioid Streaks; Peau d'Orange; Grönblad-Stranberg Disease (Pseudoxanthoma Elasticum)
Keywords: ABCC6; Pseudoxanthoma elasticum; PXE; Angioid streaks; Peau d'orange; Grönblad-Strandberg Syndrome
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Angioid Streaks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pseudoxanthoma elasticum (PXE): Genetically confirmed PXE patients
- Controls: Healthy eyes of control participants

SUMMARY:
This monocentric clinical observational study at the University Eye Hospital Bonn investigates the natural history and structural consequences of a diseased Bruch's membrane (BrM) in Pseudoxanthoma elasticum (PXE). The study includes four main objectives:

1. Direct Bruch's Membrane Alterations: Longitudinal analysis of BrM reflectivity using high-resolution OCT to assess correlations with disease progression
2. Choriocapillaris Flow Deficits: Evaluation of choriocapillaris (CC) perfusion in relation to BrM calcification, aiming to clarify whether CC deficits precede or result from BrM changes
3. Retinal Atrophy Progression: Monitoring the development and expansion of retinal atrophic areas over two years, including correlations with specific features like reticular pseudodrusen and hyperreflective spots
4. Genotype-Phenotype Correlation: Analysis of different ABCC6 gene mutations to identify correlations with imaging features and disease severity, potentially guiding future personalized therapeutic strategies

The study will recruit 100 PXE patients and 100 controls, with data collection over 10 years. It involves non-invasive imaging and blood sampling. No direct benefit is expected for participants, but the findings may inform future clinical trials and improve patient counseling.

ELIGIBILITY:
Inclusion Criteria for PXE cohort:

* PXE based on the criteria of Plomp et al.
* Clear ocular media
* Ability to perform the tasks of the study protocol (i.e., holding the head still for image aquisition)

Exclusion Criteria:

* Any confounding ocular disease not associated with PXE
* Systemic diseases hindering the study examinations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: PXE patients will be recruited from the dedicated PXE clinic in Bonn, Germany and is open for any PXE patient (external clinics) that desire to participate.
  We will also present the study at the Annual meeting of the German PXE patient organization and with PXE international, the largest patient organization worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Eccentricity of 'Peau d'orange' over 2 years | 2 years
  'Peau d'orange' will be measured in en-face imaging [mm2]

SECONDARY OUTCOMES:
Bruch's Membrane changes on High-Resolution Optical coherence tomography (OCT) | 2 years
  Bruch's membrane will be qualitatively graded on High resolution OCT (integrity, breaks, ...)
Choriocapillaris flow voids on Optical Coherence Tomography Angiography (OCT-A) | 2 years
  Choriocapillaris degeneration will be evaluated on OCT-Angiography, i.e. percent (%) of flow voids, progression over 2 years
Angioid Streak Length on Fundus Photography and Infrared Reflectance Imaging | 2 years
  Angioid Streaks will be measured manually with the unit [mm]

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University Hospital Bonn, Germany, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided